CLINICAL TRIAL: NCT05001646
Title: Clinical and Molecular Impact of In-home Resonance-based Electromagnetic Field Protection Device Usage in Healthy Individuals
Brief Title: Electromagnetic Field Protection Device Use Impact in Healthy Volunteers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TruDiagnostic (Industry)
Collaborators: Blushield USA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALT-BS-001
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Aging; Aging Well

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-home EMF protection device (Experimental)
  Interventions: Device: In-home resonance-based electromagnetic field protection device

INTERVENTIONS:
Device: In-home resonance-based electromagnetic field protection device — Participants will have an in-home EMF protection device

SUMMARY:
This is a prospective, single group, self-controlled study to evaluate the clinical and molecular impact of continuous in-home resonance-based electromagnetic field (EMF) protection device usage in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Any sex, gender orientation, and ethnicity
* Between ages 30 and 70
* Must be willing and able to participate in venipuncture, health history and clinical assessments, passive monitoring (Oura ring), and continuous in-home Blushield device usage

Exclusion Criteria:

* Significant change in diagnosis and/or treatment of major illness or injury within 2 years prior to screening, e.g., diabetes, cancer, cardiovascular disease, psychiatric condition 2. Any ongoing immune system concerns or immunodeficiency disease
* History of any viral illness in preceding year
* Body mass index (BMI) > 35 kg/m2
* Presence of active infection
* Any other illness, disorder, alcohol or chemical dependence that in the opinion of investigators would render study participation unsuitable
* Unable or unwilling to provide required biological sample
* Unable or unwilling to avoid pregnancy during study period

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Testing | Change from baseline to 12 weeks

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hernandez-Segura A, Nehme J, Demaria M. Hallmarks of Cellular Senescence. Trends Cell Biol. 2018 Jun;28(6):436-453. doi: 10.1016/j.tcb.2018.02.001. Epub 2018 Feb 21. PMID 29477613
- [Background] Karipidis K, Mate R, Urban D, Tinker R, Wood A. 5G mobile networks and health-a state-of-the-science review of the research into low-level RF fields above 6 GHz. J Expo Sci Environ Epidemiol. 2021 Jul;31(4):585-605. doi: 10.1038/s41370-021-00297-6. Epub 2021 Mar 16. PMID 33727687
- [Background] Kohli J, Wang B, Brandenburg SM, Basisty N, Evangelou K, Varela-Eirin M, Campisi J, Schilling B, Gorgoulis V, Demaria M. Algorithmic assessment of cellular senescence in experimental and clinical specimens. Nat Protoc. 2021 May;16(5):2471-2498. doi: 10.1038/s41596-021-00505-5. Epub 2021 Apr 28. PMID 33911261